CLINICAL TRIAL: NCT05004766
Title: Effects of Virtual Reality Application on Pain Reduction and Cerebral Blood Flow in Robot-Assisted Gait Training in Burn Patients : Pilot Study
Brief Title: Effects of Virtual Reality Application on Pain Reduction and Cerebral Blood Flow in Robot Training in Burn Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangangSHH-12
Record Dates: First submitted 2021-07-29; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Burns; Pain; Virtual Reality
Keywords: burns; pain; virtual reality; robot assisted hait training; functional near infrared spectroscopy
MeSH Terms: conditions — Burns; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality apply (Experimental): Using the VR system during robot training, the auditory stimulation of VR was applied along with the image of walking of a forest road or coastal road at the same speed as the robot walking speed. The VR programs are a composition of scenic beaty with sounds of nature. Each program is a blend of scenes such as the ocean, desert, forest, flowers, waterfalls, and wildlife.
  Interventions: Other: Robot assisted gait training with virtual reality
- control condition (No Intervention): Each patient participated in the control condition, during which he or she performed RAGT with no distraction for the same amount of time spent doing therapy in VR.

INTERVENTIONS:
Other: Robot assisted gait training with virtual reality — Using the VR system during robot training, the auditory stimulation of VR was applied along with the image of walking of a forest road or coastal road at the same speed as the robot walking speed. The VR programs are a composition of scenic beaty with sounds of nature. Each program is a blend of scenes such as the ocean, desert, forest, flowers, waterfalls, and wildlife.
  Arms: virtual reality apply

SUMMARY:
The purpose of this study is to determine whether the application of virtual reality (VR) is effective in reducing training pain in robot-assisted gait training (RAGT) in patients with lower extremity burn. The investigators investigated through an analysis of the activation status over time in the prefrontal cortex using functional near-infrared spectroscopy (NIRS).

DETAILED DESCRIPTION:
Burn injuries and their treatment are considered to be among the most painful a person can endure. Therefore, new modalities that prove effective with burn patients are expected to improve clinical outcomes when applied to painful therapies. The purpose of this study is to determine whether the application of virtual reality (VR) is effective in reducing training pain in robot-assisted gait training (RAGT) in patients with lower extremity burn. The investigators investigated through an analysis of the activation status over time in the prefrontal cortex using functional near-infrared spectroscopy (NIRS). RAGT was performed 10 times for 2 weeks from Monday to Friday, and the cerebral blood flow measurement using NIRS was measured 3 times each while applying or not applying VR for 30 minutes as long as the RAGT is in progress. The VR program provided non-immersive VR walking along a forest path or a coastal path according to the walking speed while the RAGT was in progress. For each physical therapy session, each patient spent equal amounts of time in VR and in the control condition (without VR). The average of oxy-Hb and deoxy-Hb of each session was measured for 10 days. In the prefrontal cortex, the levels of hemoglobin (Hb) were measured using the fNIRS measurement system. Average values of both oxy-Hb and deoxy-Hb were calculated at four stages : temporal delay time with RAGT, RAGT without VR, temporal delay time with VR, RAGT with VR. Before training, all patients verbally rated their most severe pain during physical training as a score of 5 or higher on a visual analog scale (VAS) of 0 to 10, where 0 presents " no pain at all" and 10 presents " worst pain". Pain, the primary dependent variable, was measured immediately after each experimental treatment. Patient rated (1) their worst pain (no pain to worst pain), and (2) their average pain ( no pain or worst pain).

ELIGIBILITY:
Inclusion Criteria:

* partial-to-full-thickness burns that had spontaneously healed or required skin grafting
* all patients rated their most severe pain during robot assisted gati training (RAGT) as a score 5 or higher on a visual analog scale of 0 to 10, where 0 represents no pain at all, and 10 represents worst pain.
* 1 ≤ functional ambulation category (FAC) score ≤ 3

Exclusion Criteria:

* patients with history of brain injury
* cognitive disorders, intellectual impairment before burn injury
* problems with weight bearing due to unstable fractures
* body weight ≥100 kg
* severe fixed contracture
* skin disorders that could be worsened by RAGT and conventional rehabilitation

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-08-20 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
worst pain score | baseline
  0 presents " no pain at all" and 10 presents "worst pain".
worst pain score | after 10 days training
  0 presents " no pain at all" and 10 presents "worst pain".

SECONDARY OUTCOMES:
average pain | baseline
  0 presents " no pain at all" and 10 presents "worst pain".
average pain | after 10 days training
  0 presents " no pain at all" and 10 presents "worst pain".
cerebral blood flow of prefrontal cortex | baseline
  oxygenated hemoglobin (HbO2) and deoxygenated hemoglobin (HbR) concentration will be measured using an fNIRS device (NIRSIT®; OBELAB Inc., Seoul, Korea) while the participants is training with exoskeleton robot.
cerebral blood flow of prefrontal cortex | after 10 days training
  oxygenated hemoglobin (HbO2) and deoxygenated hemoglobin (HbR) concentration will be measured using an fNIRS device (NIRSIT®; OBELAB Inc., Seoul, Korea) while the participants is training with exoskeleton robot.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joo SY, Cho YS, Lee SY, Seok H, Seo CH. Effects of Virtual Reality-Based Rehabilitation on Burned Hands: A Prospective, Randomized, Single-Blind Study. J Clin Med. 2020 Mar 9;9(3):731. doi: 10.3390/jcm9030731. PMID 32182742
- [Background] Yucel MA, Aasted CM, Petkov MP, Borsook D, Boas DA, Becerra L. Specificity of hemodynamic brain responses to painful stimuli: a functional near-infrared spectroscopy study. Sci Rep. 2015 Mar 30;5:9469. doi: 10.1038/srep09469. PMID 25820289